CLINICAL TRIAL: NCT00102609
Title: A Phase I Study to Determine the Dose of the Combination of Yondelis and Doxorubicin for Which Neutropenia is Manageable With the Support of Granulocyte-Colony Stimulation Factor in Subjects With Recurrent or Persistent Soft Tissue Sarcoma
Brief Title: A Safety Study Utilizing Yondelis and Doxorubicin in Patients With a Type of Cancer Called Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry); PharmaMar S.A.U. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003250; ET743SAR1001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2005-01-31; First posted 2005-02-01 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Soft Tissue Sarcoma; Sarcoma; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms
Keywords: Doxorubicin; Adriamycin; Trabectedin; Yondelis; Ecteinascidin 743; Filgrastim, Antineoplastic; Antineoplastic Agents; Pharmacologic Actions; Alkylating Agents
MeSH Terms: conditions — Sarcoma; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms | interventions — Doxorubicin; Trabectedin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trabectedin and doxorubicin (Experimental): Doxorubicin (50 to 75 mg/m2) administered intravenously on Day 1 followed by trabectedin (0.9 to 1.3 mg/m2) administered intravenously on Day 1 every 3 weeks for up to 6 cycles. Dexamethasone 20 mg administered intravenously will be given within 1 hour before the start of doxorubicin. Patients may receive filgrastim for unmanageable neutropenia.
  Interventions: Drug: Doxorubicin; Drug: Trabectedin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 50 to 75 mg/m2 administered intravenously on Day 1
Drug: Trabectedin — Trabectedin 0.9 to 1.3 mg/m2 administered intravenously on Day 1 every 3 weeks for up to 6 cycles
Drug: Dexamethasone — Dexamethasone 20 mg administered intravenously within 1 hour before the start of doxorubicin

SUMMARY:
The purpose of the study is to determine the dose of the combination of trabectedin (Yondelis) and Doxorubicin for which neutropenia (low white blood cell counts) could be managed with filgrastim (a Granulocyte-Colony Stimulation Factor that is used to help control neutropenia) in patients with a type of cancer called soft tissue sarcoma.

DETAILED DESCRIPTION:
This is a multicenter, open-label (identity of the assigned study treatments will be known to patients and study staff) study to determine the dose of the combination of trabectedin (Yondelis) and Doxorubicin for which the neutropenia (low white blood cell counts) is manageable with the use of filgrastim (an agent used to manage neutropenia) and associated with clinically acceptable number of side effects severe enough to continuation of treatment in patients with recurrent or persistent soft tissue sarcoma (STS, a malignant tumor that attacks the body's infrastructure of fat, muscles, nerves, joints, blood vessels, or deep skin tissues). Patients will be enrolled in the study after all study-specific entry criteria are met and informed consent is obtained. Patients will be required to attend regular clinic visits to receive study medication and have their status monitored. A detailed explanation can be provided by the study physician (Investigator) conducting this study. Doxorubicin (50 to 75 mg/m2) will be given as a 10-15 minute intravenous (i.v.) infusion on Day 1 via a central venous catheter which is a tube placed into a large vein. Trabectedin (0.9 to 1.3 mg/m2) will be given as a 3 hour i.v. infusion, immediately following the administration of doxorubicin. Dexamethasone 20 mg will be given within 1 hour before the start of each doxorubicin i.v. infusion and filgrastim will be administered according to manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of soft tissue sarcoma, recurrent or persistent
* Signed informed consent obtained for all patients before performing any study-related procedures

Exclusion Criteria:

* Patients treated with more than 1 prior chemotherapy regimen (including adjuvant (or other additional) therapy)
* Previous exposure to anthracyclines (a class of drugs used in cancer chemotherapy, example is Doxorubicin) or trabectedin
* Less than 4 weeks since radiation therapy
* Known metastases (spread) of cancer to the central nervous system
* Other ongoing serious illness present at the time of enrollment as determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety | Up to approximately 19 weeks (six 3-week treatment cycles+30 day safety follow up)

SECONDARY OUTCOMES:
The number of patients with clinically relevant changes in clinically laboratory tests | Up to approximately19 weeks (six 3-week treatment cycles+30 day safety follow up)
Number of patients with neutropenia | Up to approximately19 weeks (six 3-week treatment cycles+30 day safety follow up)
Plasma concentrations of trabectedin (Yondelis) | During the first 3 weeks of treatment
Plasma concentrations of Doxorubicin | During the first 3 weeks of treatment
Plasma concentrations of Doxorubicinol | During the first 3 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, LLC Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research and Development, LLC